CLINICAL TRIAL: NCT00427609
Title: Efficacy of Bicillin LA for the Treatment of Chronic, Plaque-type Psoriasis Unresponsive to Topical Medications.
Brief Title: Bicillin L-A vs Placebo for the Treatment of Chronic, Plaque-Type Psoriasis Unresponsive to Topical Medications
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough enrollees to obtain a valid conclusion
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8389
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Psoriasis
Keywords: Treatment; Psoriasis; efficacy; Bicillin
MeSH Terms: conditions — Psoriasis | interventions — Penicillin G Benzathine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Bicillin L-A
- 2 (Active Comparator)
  Interventions: Drug: Bicillin L-A

INTERVENTIONS:
Drug: Bicillin L-A — Bicillin L-A administered intramusculary in a dose of 2.4 million units every three weeks or normal saline injection administered intramusculary in a dose of 3 cc every three weeks

SUMMARY:
The purpose of this study is to determine the efficacy for Bicillin L-A, administered intramuscularly in a dose of 2.4 million units every three (3) weeks, for the treatment of chronic, plaque-type psoriasis unresponsive to topical medications or when other systemic therapies are contraindicated.

DETAILED DESCRIPTION:
Psoriasis is a chronic, inflammatory skin disorder most commonly manifested by well-demarcated, erythematous and/or scaling plaques on the elbows, knees, scalp, and trunk. Psoriasis is a common disease with overall incidence of 1-3% of the general population. The estimated prevalence varies from 1-2%. There is significant geographical variability with the lowest incidence of the disease around the equator and increasing towards the poles.

Psoriasis is now considered an autoimmune disease mediated by activated T-cells, releasing proinflammatory cytokines, predominately TNF-a and IFN-y. The key role for T-cells in the pathogenesis of psoriasis was supported by reported beneficial effects of specific T cell targeted therapies including cyclosporin A and certain recently marketed immune response modifiers.

While disease pathogenesis is still not completely understood, the factors that may trigger or worsen psoriasis have been systematically studied and well described in the medical literature. Psychological stress, mechanical trauma to the skin, certain medications and Streptococcus strains are the most common disease triggers.

It was first reported in 1916 that the onset of psoriasis is often preceded by throat infections with hemolytic streptococci and the role of M-protein positive beta hemolytic streptococci in triggering guttate psoriasis has been confirmed in subsequent studies. Exacerbation of chronic plaque type psoriasis has been reported in association with tonsillitis in retrospective studies. Moreover, high frequency of remission after tonsillectomy or antibiotic treatment has been documented.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age (with onset before age 40)
* Presence of chronic plaque type psoriasis unresponsive to treatment with topical preparations and extensive enough to consider appropriateness of systemic therapy
* Guttate forms of psoriasis
* Non-responsive to treatment or worsening of the pre-existing psoriasis
* With the exception of their skin disease , in good general state of health based on a complete medical history, blood test and urine analysis.
* Females must have negative urine pregnancy test and willing to take additional measures to keep from becoming pregnant during the course of the study
* No systemic prescription medication to control psoriasis within past 30 days
* Free of any topical antipsoriatic preparation for the duration of the study with the exception of emollients and moisturizers

Exclusion Criteria:

* Pustular forms of psoriasis, either localized or generalized
* Generalized Erythrodermic psoriasis
* Only palmoplantar psoriasis
* Only scalp psoriasis
* Only nail psoriasis
* Only inverse psoriasis
* Diabetes or impaired glucose tolerance
* History of recurrent yeast infections
* History of hypersensitivity to Penicillin
* History of severe adverse drug reactions
* Pregnancy
* Lactation
* HIV/AIDS
* History of renal disease
* History of liver disease
* History or presence of alcohol and/or drug dependence or abuse
* History of significant psychiatric illness
* History of allergy, asthma, allergic rhinitis, or urticaria subjects in other research trials, at least 30 days prior to the beginning of this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
A reduction of an individual's PASI by 75% after five (5) treatments of the active drug (Bicillin L-A). To demonstrate benefit comparable to the currently available biologicals, the response rate of Bicillin L-A must be at least 40% | One year

CONTACTS AND LOCATIONS:
Overall Officials: Elias Rosenberg, MD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States